CLINICAL TRIAL: NCT00471952
Title: Maxalt 10mg Plus Caffeine 75mg in the Acute Treatment of Migraine Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Diamond Headache Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DHC 09
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Migraine With Aura; Migraine Without Aura
Keywords: Migraine
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura; Migraine Disorders | interventions — rizatriptan; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Maxalt 10mg with Caffeine 75mg
  Interventions: Drug: Maxalt 10mg MLT plus Caffeine 75mg
- 2 (Active Comparator): Maxalt 10mg plus Placebo
  Interventions: Drug: Maxalt 10mg MLT plus Placebo
- 3 (Placebo Comparator): Double placebo
  Interventions: Drug: Placebo + Placebo

INTERVENTIONS:
Drug: Maxalt 10mg MLT plus Caffeine 75mg — One migraine attack will be treated
  Arms: 1
Drug: Maxalt 10mg MLT plus Placebo — One migraine attack will be treated with Maxalt 10mg plus placebo
  Arms: 2
Drug: Placebo + Placebo — One migraine attack will be treated with double placebo
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the effect of rizatriptan, alone or combined with caffeine for treating acute attacks of migraine.

Each subject will have 3 months to treat 3 acute migraine headache attacks. Each subject will be dispensed one box containing 3 packets of study medication labeled for Headache #1, Headache #2, or Headache #3. Each packet wil contain either Maxalt 10mg MLT or a Maxalt placebo (sugar pill), and a capsule containing either caffeine 75mg or a capsule containing placebo (sugar).

One headache will be treated with a combination of Maxalt 10mg MLT and caffeine.

Another headache will be treated with a combination of Maxalt 10mg MLT and a capsule containing placebo.

A third headache will be treated with just placebo.

Neither the subject, the study coordinator, or your study doctor will know in which order you will receive the three different treatments. This information is available in case of emergency.

DETAILED DESCRIPTION:
Oral Maxalt has an extensive record of providing relief of acute migraine headache with 2 hours in the vast majority of patients, especially when undertaken as an early intervention strategy. Caffeine has been demonstrated to have analgesic effects in patients treating tension type headache and is found as part of a combination including aspirin and acetaminophen as a treatment for acute migraine headache.

The mechanism by which Maxalt relieves migraine headache is believed to be through action on 5HT1B/1D receptors both on blood vessels as well as centrally. Caffeine may have effects on relief of migraine through modifying norepinephrine related mechanisms which have been suggested through clinical research. Patients commonly report that they may obtain partial or complete relief of their migraines by consuming the modest amounts of caffeine found in a cup of coffee. this is estimated to be approximately 100mg per cup. The analgesic effects of caffeine appear to be most significant in the first 3 hours after ingestion. Recent work suggests that intervention in migraine when the pain is still mild and has not persisted for a prolonged duration may increase the likelihood of complete migraine response. Therefore, the combination of the two agents with activity in migraine that work early in the migraine process, have good tolerability at the proposed doses and working via different mechanism may increase the likelihood of patients achieving better response with their migraine treatment than that which is currently available.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-65 years of age
* Diagnosis of migraine with or without aura
* 1 year history of migraine with 1-6 migraine attacks per month in the the three months prior to screening
* Medication for migraine prevention with a stable dose for at least 1 month prior to screening
* Has successfully treated a migraine attack with a triptan medication

Exclusion Criteria:

* Confirmed or suspected ischemic heart disease
* History of congenital heart disease
* History of cerebrovascular disease, including stroke
* History of ischemic abdominal disease
* Uncontrolled hypertension
* History of epilepsy
* History of basilar or hemiplegic migraine
* Impaired hepatic or renal function
* Greater than 15 headache days per month
* Subjects on an MAOI
* Subjects taking and ergotamine, or ergot containing preventive medication
* Subject is pregnant, trying to become pregnant or breast feeing
* Evidence of alcohol or substance abuse in the last year
* History of caffeine withdrawal headache
* Consumes more than 275 mg of caffeine on daily basis from dietary and medication sources
* Taking propanolol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The comparative percentage of migraine attacks that produce pain free response at 2 hours in the Maxalt 10mg MLT plus caffeine 75mg arm versus the Maxalt 10mg MLT plus placebo caffeine versus double placebo. | 2 hours

SECONDARY OUTCOMES:
The comparative percentage of attacks that produce pain relief at 2 hours. | 2 hours
The comparative percentage of attacks that produce a pain free response and do not require re-treatment during the subsequent 24 hours and are not associated with headache pain recurrence. | 24 hours
The comparative percentage of resolution of associated symptoms of migraine present at the time of treatment as well as achieving a pain free response within 2 hours with each of the treatments. | 2 hours
The comparative number of patients reporting adverse effects to study medication, the type of adverse events reported and the percentage of attacks that are associated with the adverse effect. | 24 hours
Patient global evaluation for each of the treatments | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Freitag, DO, Principal Investigator — Diamond Headache Clinic
Locations (1):
- Diamond Headache Clinic, Chicago, Illinois, United States